CLINICAL TRIAL: NCT03948490
Title: Rehabilitation and Longitudinal Follow-up of Cognition in Adult Lower Grade Gliomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tilburg University (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19103; NCI-2019-03245 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-03

CONDITIONS: Low-grade Glioma
Keywords: cognitive impairment; quality of life
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Arm 1 Cohort 1: Interventional arm/In-person rehab (CLOSED) (Other): The in-person cognitive rehabilitation will focus on the application of evidenced based strategies recommended as practice guidelines by the American Congress of Rehabilitation Medicine Cognitive Rehabilitation Task Force (ACRM-CR). The treatment occurs in two stages 1) comprehensive neuropsychological assessment and rehabilitation planning and 2) implementation of treatment planning.
  n = 20 patients
  Interventions: Behavioral: In-person cognitive rehabilitation
- Arm 1 Cohort 2: Interventional arm/ReMind iPad app (CLOSED) (Experimental): The ReMind iPad-based cognitive rehabilitation was developed with collaborators at Tilburg University, The Netherlands, and is an evidence-based program to improve attention and memory through (1) cognitive training and (2) teaching compensatory skills in patients with brain tumors. Brain plasticity-based computerized cognitive training is a newly developing field of therapeutics for neurological and psychiatric disorders that uses frequent game-like training sessions to drive improvements in cognitive functions.
  n = 20 patients
  Interventions: Device: ReMind iPad app
- Arm 1 Cohort 3: Interventional arm/Healthy SMS texting (CLOSED) (Experimental): The mobile phone texting intervention was developed with collaborators at Zuckerberg San Francisco General Hospital and is currently being studied in individuals with depression and traumatic brain injury. Participants receive a daily message sent at a random time (within their chosen timeframe(s); e.g. 9am-9pm). Messages will focus on patient-based education-focused health-related quality of life and cognitive education such as internal and external cognitive compensatory strategy training, fatigue management, and coping skills.
  n = 20 patients
  Interventions: Device: Healthy SMS texting
- Arm 2 Cohort 4: Longitudinal arm/Upfront radiation (No Intervention): Patients will undergo longitudinal global cognitive and HRQOL assessments at baseline prior to surgery, after surgery, 3 months after surgery and every 6 months for 3 years. Clinical data will be collected at the time of each assessment. This will include changes in serial imaging e.g. in T2 tumor volume, DTI scalar quantification, resting-state fMRI connectivity n = 50 patients
- Arm 1 Cohort 5: Longitudinal arm/No upfront radiation (No Intervention): Patients will undergo longitudinal global cognitive and HRQOL assessments at baseline prior to surgery, after surgery, 3 months after surgery and every 6 months for 3 years. Clinical data will be collected at the time of each assessment. This will include changes in serial imaging e.g. in T2 tumor volume, DTI scalar quantification, resting-state fMRI connectivity n = 50 patients
- Arm 1 Cohort 1A: Telehealth Cognitive Rehabilitation (Other): The telehealth cognitive rehabilitation will take place over secure UCSF Zoom. It will focus on the application of evidenced based strategies recommended as practice guidelines by the American Congress of Rehabilitation Medicine Cognitive Rehabilitation Task Force (ACRM-CR). The treatment occurs in two stages 1) comprehensive neuropsychological assessment and rehabilitation planning and 2) implementation of treatment planning. During treatment implementation, patients acquire, apply, and adapt evidenced based strategies based on neuropsychological testing and conjointly developed treatment planning goals.
  N=20
  Interventions: Behavioral: Telehealth cognitive rehabilitation

INTERVENTIONS:
Device: ReMind iPad app — Evidence-based program to improve attention and memory through (1) cognitive training and (2) teaching compensatory skills in patients with brain tumors.
  Arms: Arm 1 Cohort 2: Interventional arm/ReMind iPad app (CLOSED)
Device: Healthy SMS texting — Participants receive a daily message sent at a random time (within their chosen timeframe(s); e.g. 9am-9pm). Messages will focus on patient-based education-focused health-related quality of life and cognitive education such as internal and external cognitive compensatory strategy training, fatigue management, and coping skills.
  Arms: Arm 1 Cohort 3: Interventional arm/Healthy SMS texting (CLOSED)
Behavioral: In-person cognitive rehabilitation — The in-person cognitive rehabilitation will focus on the application of evidenced based strategies recommended as practice guidelines by the American Congress of Rehabilitation Medicine Cognitive Rehabilitation Task Force (ACRM-CR). The treatment occurs in two stages 1) comprehensive neuropsychological assessment and rehabilitation planning and 2) implementation of treatment planning.
  Arms: Arm 1 Cohort 1: Interventional arm/In-person rehab (CLOSED)
Behavioral: Telehealth cognitive rehabilitation — The telehealth cognitive rehabilitation will take place over secure UCSF Zoom. It will focus on the application of evidenced based strategies recommended as practice guidelines by the American Congress of Rehabilitation Medicine Cognitive Rehabilitation Task Force (ACRM-CR). The treatment occurs in two stages 1) comprehensive neuropsychological assessment and rehabilitation planning and 2) implementation of treatment planning
  Arms: Arm 1 Cohort 1A: Telehealth Cognitive Rehabilitation

SUMMARY:
Patients with glial brain tumors have increasingly improved outcomes, with median survival of 5-15 years. However, the treatments, including surgery, radiation, and chemotherapy, often lead to impaired attention, working memory, and other cognitive functions. These cognitive deficits frequently have significant impact on patient quality of life. Although currently, there is no established standard of care to treat cognitive deficits in brain tumor patients, standard cognitive rehabilitative treatments have been developed for those with traumatic brain injury and stroke. However, the feasibility and efficacy of these cognitive treatments in individuals with brain tumors remains unclear.

DETAILED DESCRIPTION:
This trial studies how well cognitive rehabilitation therapy works in improving cognitive function in patients with lower grade gliomas. Patients with low grade gliomas frequently have symptoms of cognitive impairment, such as difficulty with short term memory and processing information, that impacts their daily lives. The ReMind application (app) is an iPad app developed for cognitive rehabilitation for patients. The healthy texting platform was developed to help patients with depression and cognitive difficulty to provide education and track their mood. Methods of cognitive rehabilitation therapy such as in person cognitive rehabilitation, computerized cognitive rehabilitation, and healthy text messaging may help improve cognition and quality of life in patient with low grade gliomas.

PRIMARY OBJECTIVES:

* Assess feasibility of each interventional arm independently (Arm 1)
* Detect a decline of >= 1.5 standard deviation (SD) from baseline on the Wechsler Adult Intelligence Scale (WAIS)- IV Working Memory Score or Hopkins Verbal Learning Test (HVLT) during the 36 month follow-up after surgery. (Arm 2)

SECONDARY OBJECTIVES:

* Measure changes in cognition at post-intervention and follow-up for each cohort - cohort 1 in-person; cohort 1A telehealth; cohort 2 ReMind; and cohort 3 short message service (SMS) texting - at 3 months and 6 months post-intervention. (Arm 1)
* Measure changes in health related quality of life (HRQOL) at post-intervention and follow-up for each cohort - cohort 1 in-person; cohort 2 ReMind; and cohort 3 SMS texting - as captured by Patient Reported Outcomes Measurement Information System-quality of life (PROMIS-QOL) - at 3 months and 6 months post-intervention. (Arm 1)
* Assess relationships between cognitive changes and clinical factors (molecular subtype, age, tumor location, treatment, and radiation fields when appropriate). (Arm 2)
* Assess relationships between cognitive changes and serial magnetic resonance (MR) imaging (T2 and contrast-enhancing tumor volume, diffusion tensor imaging (DTI) scalar quantification, structural connectivity, resting-state functional magnetic resonance imaging (fMRI) connectivity). (Arm 2)
* Assess relationships between HRQOL and cognitive changes. (Arm 2)

EXPLORATORY OBJECTIVES:

* Assess relationships between cognitive and HRQOL. (Arm 1)
* Assess relationships between cognitive changes and clinical factors (molecular subtype, age, tumor location, and radiation fields when appropriate). (Arm 1)
* Assess relationships between HRQOL changes and clinical factors (molecular subtype, age, tumor location, and radiation fields when appropriate). (Arm 1)
* Assess relationships between cognitive changes and serial MR imaging (T2 and contrast-enhancing tumor volume, DTI scalar quantification, structural connectivity, resting-state fMRI connectivity). (Arm 1)
* Identify predictive power of tumor characteristics (tumor volume, location, molecular characteristics), patient characteristics (extent of resection, treatment, and radiation fields when appropriate), imaging characteristics (e.g. fMRI, DTI changes), and decline in cognition or HRQOL. (Arm 2)

OUTLINE:

Patients are invited to participant in Cohort 1A. Patients unable to participant in Cohort 1A are randomized to Cohort 2 or Cohort 3.

ARM 1:

* COHORT 1 (CLOSED): Patients receive standard in-person cognitive rehabilitation sessions with a neuropsychologist every 2 weeks over 1 hour each for 12 weeks.
* COHORT 1A: Patients receive telehealth cognitive rehabilitation with University of California, San Francisco (UCSF) Zoom visits with a neuropsychologist who specializes in brain tumors over 60 minutes every 2 weeks for 3 months.
* COHORT 2 (CLOSED): Patients receive computerized cognitive rehabilitation using the ReMind app over 3 hours per week for 12 weeks.
* COHORT 3 (CLOSED): Patients receive healthy text messages daily at random points during the week (Monday - Friday) for 12 weeks.

ARM 2:

* COHORT 4: Patients who receive radiation after surgery, undergo longitudinal cognitive and health related quality of life assessments prior to surgery, prior to start of radiation, at 4-6 week after radiation, 6 and 12 months after surgery, and then every 6 months for 36 months after surgery.
* COHORT 5: Patients who do not receive radiation after surgery, undergo longitudinal cognitive and health related quality of life assessments prior to surgery, within 1 month after surgery, 2-4 months after surgery, 6 and 12 months after surgery, and then every 6 months for 36 months after surgery.

After completion of study, patients in cohorts 1-3 are followed up at 3 and 9 months.

ELIGIBILITY:
Arm 1:

Inclusion Criteria:

* Histologically confirmed low grade supratentorial primary brain tumor
* >= 18 years old
* Life expectancy > 12 weeks
* Karnofsky performance status (KPS) >= 70
* Must speak and be able to read English fluently
* Must have access to the internet
* Must have text enabled cellphone
* Must be receiving MRI scans at University of California, San Francisco (UCSF)
* Must be clinically stable and off treatment (e.g. radiation or chemotherapy) for ≥ 3 months
* Must be >= 6 months from craniotomy
* Must have subjective complaints of cognitive deficits
* Must have adequate seizure control and be on a stable, or decreasing, dose of anti-epileptics
* Must score <= 1 SD below normal on ≥ 2 or more domains of baseline neuropsychological assessments

Exclusion Criteria:

* Diagnosis or evidence of any of the following:
* • Glioblastoma
* • Extra-axial disease (i.e. meningioma)
* • Infra-tentorial disease
* Are not able to comply with study and/or follow-up procedures
* Are unable to complete or score >= 3 cognitive tests at baseline, which is indicative that patients would be unable to complete the cognitive rehabilitation interventions
* Are acutely suicidal, psychotic, and/or gravely disabled.
* Patients who, based on the neuropsychologist's opinion, are unable to participate in cognitive testing and/or cognitive rehab secondary to significant neurologic deficit

Arm 2:

Inclusion Criteria:

* Have a presumed low grade primary brain tumor and either be undergoing definitive surgery or have had surgical resection within the last 4 months.
* Prior surgery is allowed if they have not received additional tumor directed treatment.
* >= 18 years old
* Must speak and be able to read English fluently.
* Plan to continue to care in neuro-oncology at UCSF
* Must be receiving MRI scans.

Exclusion Criteria:

* Diagnosis or evidence of any of the following:
* • Glioblastoma
* • Extra-axial disease (i.e. meningioma)
* Are not able to comply with study and/or follow-up procedures
* Have acute psychiatric issues (suicidality, active psychosis, gravely disabled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who complete all of the intervention exercises for each cohort (Arm 1) | 9 months
  The intervention will be considered feasible for a larger-scale efficacy study if greater than 80% of the subjects complete the intervention. Patients will be replaced if they drop out of the intervention (either by declining their first follow-up visit for Cohort 1 in-person rehab; declining to participate in the Cohort 2 ReMind intervention; or by texting the word "STOP" in the Cohort 3 short message service (SMS) texting intervention)) within the first 14 days. These patients will be replaced. All other patients will be evaluable for feasibility if they remain in the Cohort past the first 14 days of the intervention
Number of participants who show a decline of >= 1.5 SD from baseline on the Wechsler Adult Intelligence Scale IV (WAIS-IV) Working Memory Score or Hopkins Verbal Learning Test (HVLT) (Arm 2) | 3 years
  Detect a decline of greater than 1.5 standard deviation (SD) compared to baseline on WAIS-IV Working Memory Score or HVLT during the 36 month follow-up after surgery

SECONDARY OUTCOMES:
Improvement of ≥1.5 SD in at least one cognitive domain at post-intervention and/or follow-up for each Cohort (Arm 1) | 9 months
  Changes in cognitive domains overtime will focus on changes in WAIS-IV Working Memory Score from baseline to post-intervention and/or follow-up within each cohort with a goal to detect the first time point at which there is at least a 1.5 standard deviation difference from baseline average
Improvement of ≥1.5 SD in health related quality of life (HRQOL) as measured by Patient-Reported Outcomes Measurement Information System (PROMIS-NeuroQOL) at post-intervention and/or follow-up for each Cohort (Arm 1) | 9 months
  Measure changes in HRQOL for each Arm 1 cohort - Cohort 1 in-person; Cohort 2 ReMind; and Cohort 3 SMS texting - as captured by Patient-Reported Outcomes Measurement Information System (PROMIS-QOL) - at post-intervention (3 months from baseline) and 6 months (9 months from baseline) post-intervention
Assess relation ships between cognitive changes and clinical factors (Arm 2) | 3 years
  Identify clinical factors (molecular subtype, age, tumor location, treatment) that correlate with ≥1.5 SD in at least one cognitive domain
Assess relationships between cognitive changes and serial magnetic resonance (MR) imaging (Arm 2) | 3 years
  Identify MR imaging characteristics (T2 FLAIR tumor volume at each imaging, T1 contrast enhancement volume at each imaging, Median, 10%, 90% apparent diffusion coefficient (ADC) and fractional anisotropy (FA) within T2 and T1 contrast tumor volumes, DTI scalar quantification and structural connectivity, Cerebral Blood Flow (CBF) within T2 and T1 contrast tumor volumes, Resting-state fMRI connectivity within the following major functional networks: default mode network, sensory/motor network, executive network, salience network, visual network and auditory network) at each time that correlate with >=1.5 SD in at least one cognitive domain.
Correlation of PROMIS-NeuroQOL scores and cognitive changes (Arm 2) | 3 years
  The changes in HRQOL as measured by PROMIS-NeuroQOL will be correlated using Spearman's rank correlation changes in >=1.5 standard deviation on at least one cognitive domain. The PROMIS-NeuroQOL is a 5 item scale which measures how much difficulty specific tasks are to complete. Item scores range from 5="None" to 1="Cannot do". The Spearman's correlation coefficient (rs) measures the strength and direction of association between two variables and can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.
Correlation between isodose lines and cognitive changes (Arm 2) | 3 years
  The isodose lines for patients who received radiation will be correlated using Spearman's rank correlation with changes in >=1.5 standard deviation on at least one cognitive domain. The Spearman's correlation coefficient (rs) measures the strength and direction of association between two variables and can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Taylor, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No